# UAB IRB Approved 01-Feb-2019 until

#### CONSENT FORM

TITLE OF RESEARCH: A Multi-level Approach to Violence Prevention among African America 08-Apr-2019

Adolescents

**UAB IRB PROTOCOL NO.:** IRB-300000551

**PRINCIPAL INVESTIGATOR:** Yu-Mei M. Schoenberger, PhD, MPH

Lori Brand Bateman, PhD

**SPONSOR:** National Institute of Minority Health and Health Disparities

### **Purpose of the Research**

We are asking you and your child to take part in a research study. The purpose of this research study is to test a youth violence prevention intervention and to understand how a multi-component intervention may influence children's behavior and well-being. The intervention combines a social and emotional learning program with a mentoring program and community improvement activities. Twenty African American boys in 6<sup>th</sup> through 8<sup>th</sup> grade (ages 11 through 14) and their caregivers will be enrolled into the study.

### **Explanation of Procedures**

If you agree to join the study, you and your child will be asked to answer questions during interviews with members of our study team, and it will take about 60 minutes. We will ask questions about what you and your child think about school and the neighborhood; relationships between you and your child; and stressful events that may happen in the home or community. You will also be asked about your child's behavior and potential consequences at school. Your answers to these questions are important to us regardless of your life experiences. This will be the first of two surveys that we ask you and your child to complete across 4 months.

Your child will be asked to attend the violence prevention intervention that will be held once a week for 2 hours over a 3 month period (12 weeks) as well as participate in up to four community improvement activities. Examples of community improvement activities include community cleaning efforts and working in the Kingston community garden. At the end of the intervention, your child will be asked to participate in a focus group to answer questions with members of our study team and it will take about 90 minutes. We will ask questions about the intervention, specific intervention skills used, outcomes of used skills, and overall thoughts and satisfaction of the program, mentoring, and community activities.

# **Risks and Discomforts**

This study involves two types of potential risks. First, some of the questions may remind you or your child of negative events or feelings (for example, being exposed to community violence or feeling depressed). Regardless of whether you decide to be in the study, you will be offered a list of phone numbers for organizations providing helpful services (for example, help in coping with stressors). Second, some of the questions included in this study involve potentially sensitive material, such as current mental health and behavior issues. There is also a risk of breach of confidentiality, but we will make every effort to protect the confidentiality of your information.

Page 1 of 3

Version Date: 1/3/19

#### **Benefits**

You may not benefit directly from taking part in this study. The information you provide will help us to better understand issues that may affect the well-being and future success of young people in the African American community.

#### **Alternatives**

Your alternative is to not participate in this study.

# Confidentiality

Information obtained about you for this study will be kept confidential to the extent allowed by law. However, research information that identifies you may be shared with people or organizations for quality assurance or data analysis, or with those responsible for ensuring compliance with laws and regulations related to research. They include:

- the UAB Institutional Review Board (IRB). An IRB is a group that reviews the study to protect the rights and welfare of research participants.
- National Institute of Minority Health and Health Disparities
- the Office for Human Research Protections (OHRP).

The information from the research may be published for scientific purposes; however, your identity will not be given out.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

### **Voluntary Participation and Withdrawal**

Whether or not you take part in this study is your choice. There will be no penalty if you decide not to be in the study. If you decide not to be in the study, you will not lose any benefits you are otherwise owed. You are free to withdraw from this research study at any time. Your choice to leave the study will not affect your relationship with the Morton Simpson Recreational Center or the University of Alabama at Birmingham.

#### **Cost of Participation**

There will be no cost to you for taking part in this study.

# **Payment for Participation in Research**

You will receive \$30 and your child will receive \$10 at the end of the interview for your time. Ask the study staff about the method of payment that will be used for this study (e.g., check, cash, gift card, direct deposit). If you need to leave before the interview is complete, we will work with you to schedule a time that is convenient for you and your child to complete the interview. If you cannot complete the interview, we will reimburse you and your child at a rate proportional to the portion of the interview that you have completed (e.g., \$10 for 1/2 completion). You will receive \$30 and your child will receive \$10 for each interview that you complete, totaling up to \$60 for caregivers and \$20 for children across 4 months.

Page 2 of 3 Version Date: 1/3/19 Your child will receive \$5 for each session that he attends, totaling up to \$60 for 12 sessions, and \$10 for each community activity (up to four), totaling up to \$40 for four community activities. In addition, if your child attends at least 9 of the 12 sessions, he will receive \$20 at the graduation ceremony. If he attends 1 to 8 of the 12 sessions, he will receive \$10 at the graduation ceremony. Your child will receive \$10 for participating in the focus group.

### **Significant New Findings**

You will be told by the study staff if new information becomes available that might affect your choice to stay in the study.

## Questions

If you have any questions, concerns, or complaints about the research, you may contact Dr. Yu-Mei Schoenberger or Dr. Lori Bateman. They will be glad to answer any of your questions. Dr. Schoenberger's number is 205-934-1724 and Dr. Bateman's number is 205-934-2924.

If you have questions about your rights as a research participant, or concerns or complaints about the research, you may contact the UAB Office of the IRB (OIRB) at (205) 934-3789 or toll free at 1-855-860-3789. Regular hours for the OIRB are 8:00a.m. to 5:00p.m. CT, Monday through Friday.

# **Legal Rights**

You are not waiving any of your legal rights by signing this informed consent document.

### **Signatures**

Your signature below indicates that you have read (or been read) the information provided above and agree to participate in this study. You will receive a copy of this signed consent form.

| Signature of Participant 14 Years of Age and Older | Date |
|----------------------------------------------------|------|
| Signature of Parent or Guardian | Date |
| Signature of Person Obtaining Consent | Date |

Version Date: 1/3/19